CLINICAL TRIAL: NCT06049030
Title: A Phase Ia/Ib Study of HS-10516 to Investigate the Safety, Tolerance, Pharmacokinetic and Efficacy in Patients With Advanced Clear Cell Renal Cell Carcinoma
Brief Title: A Study of HS-10516 in Patients With Advanced Clear Cell Renal Cell Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-10516-101
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Advanced Clear Cell Renal Cell Carcinoma; Kidney Cancer; Renal Cancer; Recurrent Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ia dose escalation (Experimental): Participants will be assigned to pre-specified dose level to identify the MTD/MAD of HS-10516.
  Interventions: Drug: HS-10516
- Phase Ib dose expansion arm (Experimental): Participants will be assigned to the recommended dose level determined in Phase Ia to evaluate the safety, pharmacokinetics and antitumor efficacy of HS-10516
  Interventions: Drug: HS-10516

INTERVENTIONS:
Drug: HS-10516 — Oral HIF-2α inhibitor

SUMMARY:
The aim of the Phase Ia portion is to identify the maximum tolerated dose or maximum acceptable dose MTD/MAD of HS-10516. The phase Ib portion will evaluate the preliminary efficacy of HS-10516 in ccRCC.

DETAILED DESCRIPTION:
This is a Phase Ia/Ib open label multicenter study of HS-10516 in Chinese patients aged 18 years or older with advanced clear cell renal cell carcinoma who have failed or are unavailable/intolerant to standard of care. HS-10516 as a single agent, is administrated orally once daily. The aim of phase Ia, a dose escalation study, is to identify the MTD/MAD of HS-10516. The goal of Phase Ib, a dose expansion study, is to evaluate the safety, pharmacokinetics and antitumor efficacy of HS-10516.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female from 18 to 75 year-old
2. Histologically confirmed locally advanced or metastasis clear cell renal cell carcinoma whose standard treatment failed or proven unavailable or intolerant
3. Has at least one non-CNS target lesion per RESIST v1.1
4. Has an Eastern Cooperative Oncology Group performance status of 0-1
5. Has a life expectancy of ≥ 12 weeks
6. Should use adequate contraceptive measures throughout the study
7. Females subject must not be pregnant at screening
8. Has the ability to understand and willingness to sign a written informed consent before the performance of the study

Exclusion Criteria:

1. Received or being received treatment as follows:

   1. Hypoxia-induced factor inhibitors
   2. Traditional Chinese medicine indicated for tumors within 2 weeks prior to the first dose of study treatment.
   3. Cytotoxic chemotherapeutic drugs, investigational drugs or other systematic anti-tumor therapies within 3 weeks before the first dose of study treatment
   4. Colony-stimulating factors (CSFs) within 4 weeks before the first dose of study treatment
   5. Local radiotherapy within 2 weeks prior to the first dose of study treatment; more than 30% of bone marrow radiotherapy or large-area irradiation within 4 weeks before the first dose of study treatment.
   6. Major surgery within 4 weeks prior to the first dose of study treatment.
2. Has a pulse oximetry reading less than 92% at screening, requires intermittent supplemental oxygen, or requires chronic supplemental oxygen
3. Has failed to recover from a ≥ grade 2 adverse event due to prior anti-tumor therapy
4. Has another malignancy or a history of another malignancy
5. Has inadequate bone marrow reserve or organ dysfunction
6. Has a clinically significant bleeding events or tendency within 1 month prior to the first dose of study treatment
7. Has severe infections within 4 weeks prior to the first dose of study treatment
8. Has digestive system diseases may influencing ADME of study drug
9. Has a history of severe hypersensitivity reaction, or proven allergic to HS-10516 or its metabolics
10. Has any disease or condition would compromise subject safety or interfere with study assessments by investigator's decision

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2024-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: MTD/MAD of HS-10516 | Approximately 2 months
  Maximum Tolerated Dose or Maximum Acceptable Dose determined by the Number of Participants with Dose Limiting Toxicity (DLT) events during the DLT monitoring period (first 35 days of dosing) in the Dose Escalation Phase
Phase Ib: Objective Response Rate (ORR) by Independent Review Committee (IRC) | Approximately 1 year
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR will be assessed by IRC.

SECONDARY OUTCOMES:
The Number of Participants with Adverse Events | Approximately 2 years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related.
Observed maximum plasma concentration (Cmax) of HS-10516 | Approximately 2 months
  Cmax will be obtained following administration of the first dose of HS-10516 during first 2 cycles.
Time to reach maximum plasma concentration (Tmax) of HS-10516 | Approximately 2 months
  Tmax will be obtained following administration of the first dose of HS-10516 during first 2 cycles.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) following the first dose of HS-10516 | Approximately 1 year
  Area under the plasma concentration versus time curve from time zero to the last sampling time when the concentration was no less than the lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
ORR by investigators | Approximately 1 year
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Disease Control Rate (DCR) | Approximately 1 year
  DCR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) or a stable disease (SD) of 8 weeks or longer based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Duration of Response (DoR) | Approximately 1 year
  DoR is defined as the time from the date of first documented CR or PR, assessed by investigator and based on RECIST v. 1.1, to the documented date of progressive disease (PD) or death, whichever occurred first.
Progression Free Survival (PFS) | Approximately 2 years
  PFS defined as the time from the date the participant started study drug to the date the participant experiences an event of disease progression or death.
Overall Survival (OS) | Approximately 2 years
  OS defined as the time from the date the participant started study drug to death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, M.D., Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: No